CLINICAL TRIAL: NCT03705923
Title: Metabolic Characterization of Subjects With Adipositas Before and After Bariatric Surgery
Brief Title: Effect of Bariatric Surgery on Brain Insulin Sensitivity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 714/2017BO1
Record Dates: First submitted 2018-08-09; First posted 2018-10-15 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bariatric surgery (Experimental): Subjects undergoing laparoscopic Roux-en-Y gastric bypass or laparoscopic sleeve gastrectomy.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — laparoscopic Roux-en-Y gastric bypass or laparoscopic sleeve gastrectomy

SUMMARY:
Adiposity is associated with prediabetes and type 2 diabetes. In very severe cases of adiposity in combination with type 2 diabetes, bariatric surgery has proven to be a successful therapy option. So far the molecular mechanisms that lead to an improvement of type 2 diabetes after bariatric surgery are not fully understood. It is planned to characterize the metabolic and neuroendocrine changes in subjects before and after bariatric surgery. One special focus of the study is brain insulin resistance, a condition known to be associated with obesity with impact on the brain and whole body metabolism.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* planned bariatric surgery (laparoscopic Roux-en-Y gastric bypass or laparoscopic sleeve gastrectomy)
* stable medication 10 weeks before begin of the study

Exclusion Criteria:

* persons who wear non-removable metal parts in or on the body.
* persons with reduced temperature sensitivity and / or increased sensitivity to heating of the body
* cardiovascular disease can not be ruled out, e.g. manifest coronary heart disease, heart failure greater than NYHA 2, previous heart attack, stroke condition
* persons with hearing impairment or increased sensitivity to loud noises
* people with claustrophobia
* minors or non-consenting subjects are also excluded
* subjects with an operation less than 3 months
* neurological and psychiatric disorders
* subjects with hemoglobin Hb <11 g / dl
* hypersensitivity to any of the substances used

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Central insulin sensitivity | Central insulin sensitivity will be assessed as change before bariatric surgery and 6 months afterwards.
  Central insulin sensitivity will be assessed by fMRI after application of nasal insulin or placebo.
Peripheral insulin sensitivity | Peripheral insulin sensitivity will be assessed by oral glucose tolerance as change before bariatric surgery and 6 months afterwards.
  Peripheral insulin sensitivity will be assessed by oral glucose tolerance test.

SECONDARY OUTCOMES:
Whole body fat distribution | Body fat distribution will be assessed by MRI prior bariatric surgery and 6 months afterwards.
  Body fat distribution will be assessed by MRI
Liver fat content | Liver fat content will be assessed by MRS prior bariatric surgery and 6 months afterwards.
  Liver fat content will be assessed by MRS
Metabolic rate | Metabolic rate will be assessed by indirect calorimetry prior bariatric surgery and 6 months afterwards.
  Metabolic rate will be assessed by indirect calorimetry
Response to food cues | Change in response to food cues will be assessed before bariatric surgery and 6 months afterwards.
  Food cues will be rated for palatability on a visual analogue scale
Trail-making test | Change in trail-making test will be assessed before bariatric surgery and 6 months afterwards.
  Trail-making test will be performed
Hopkins-verbal learning test | Change in Hopkins-verbal learning test will be assessed before bariatric surgery and 6 months afterwards.
  Hopkins-verbal learning test will be performed
Glucose tolerance | Glucose tolerance will be assessed by 75g oral glucose tolerance test prior to bariatric surgery and 6 months afterwards.
  Glucose tolerance will be assessed by 75g oral glucose tolerance test.
Insulin secretion | Insulin secretion will be assessed by insulin measurements during 75g oral glucose tolerance test prior to bariatric surgery and 6 months afterwards.
  Insulin secretion will be assessed by insulin measurements during 75g oral glucose tolerance test.
Weight loss | Weight loss before and 6 months after surgery.
  Body weight will be measured before and 6 months after surgery.

OTHER OUTCOMES:
Liver, adipose tissue and muscle specimens | At surgery
  During surgery liver, subcutaneous and visceral adipose tissue and skeletal muscle will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No